CLINICAL TRIAL: NCT05638035
Title: Effects of Obesity on Rectus Femoris Muscle Thickness, Sarcopenia, Gait and Balance in Women
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Yağmur KURALAY, physiotherapist, Kutahya Health Sciences University
Other Study IDs: DSA2022
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Sarcopenic Obesity; Sarcopenia; Obesity
MeSH Terms: conditions — Sarcopenia; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-obese women: After obtaining demographic information for women with a BMI of 18-27.9 kg/m2 for at least 6 months, Body Mass Index (BMI) will be calculated and the relationship between rectus femoris muscle thickness, sarcopenia, gait and balance will be evaluated and will be compared with obese group.
  Interventions: Diagnostic Test: Ultrasonografi, Sarcopenia measurement, Zebris
- obese women: After obtaining demographic information in women with a BMI of 30-39.9 kg/m2, Body Mass Index (BMI) will be calculated and the relationship between obesity and rectus femoris muscle thickness, sarcopenia, gait and balance will be evaluated.
  Interventions: Diagnostic Test: Ultrasonografi, Sarcopenia measurement, Zebris

INTERVENTIONS:
Diagnostic Test: Ultrasonografi, Sarcopenia measurement, Zebris — The rectus femoris muscle thickness of the participants will be performed in B mode via USG (Mindray-UMT 200,USA) with a multifrequency (7-15 MHz) linear probe and the measurement will be reported.
  TANITA for sarcopenia, hand grip strength and walking speed will be evaluated.
  Gait time-distance parameters and Static balance COP parameters (COP speed (cm/s) and COP length (cm)) will be recorded using Zebris™ FDM-2.

SUMMARY:
Research; It is a planned, non-invasive, controlled study in obese female volunteers and non-obese female volunteers. The population of the study consists of voluntarily non-obese women and obese women. Sarcopenia assets of individuals will be measured with the sarc-f questionnaire, and then muscle strength, muscle mass and physical performance tests will be measured. Then, rectus femoris muscle thickness will be measured with USG, and then walking and balance will be measured with ZEBRIS.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old and female
* Volunteering and accepting to participate in the study
* BMI 30-39.9 kg/m2 in obese women (experimental group)
* BMI 18-27.9 kg/m2 in non-obese women (control group)
* Not having cardiorespiratory, neurological, orthopedic and metabolic disorders

Exclusion Criteria:

* Being under 18 years old and male
* Having a BMI of 40.0 kg/m2 and above in obese women (experimental group)
* BMI 28.0 kg/m2 and above in non-obese women (control group)
* Having cardiorespiratory, neurological, orthopedic and metabolic disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women will be included in the study.
Study Population: The population of the research consists of voluntarily non-obese women residing in Kütahya/Center and obese women voluntarily participating in the study at Kütahya Evliya Çelebi Training and Research Hospital Physical Therapy and Rehabilitation Hospital Obesity School.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Rectus femoris muscle thickness | baseline
  Measurement of muscle thickness with ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: yagmur kuralay, Principal Investigator — kütahya health sciences university
Locations (1):
- Kütahya Health Sciences University, Kütahya, Centre, Turkey (Türkiye)

REFERENCES:
- [Background] Mueller N, Murthy S, Tainter CR, Lee J, Riddell K, Fintelmann FJ, Grabitz SD, Timm FP, Levi B, Kurth T, Eikermann M. Can Sarcopenia Quantified by Ultrasound of the Rectus Femoris Muscle Predict Adverse Outcome of Surgical Intensive Care Unit Patients as well as Frailty? A Prospective, Observational Cohort Study. Ann Surg. 2016 Dec;264(6):1116-1124. doi: 10.1097/SLA.0000000000001546. PMID 26655919
- [Background] Dutil M, Handrigan GA, Corbeil P, Cantin V, Simoneau M, Teasdale N, Hue O. The impact of obesity on balance control in community-dwelling older women. Age (Dordr). 2013 Jun;35(3):883-90. doi: 10.1007/s11357-012-9386-x. Epub 2012 Feb 10. PMID 22318311
- [Background] Ates Bulut E, Soysal P, Dokuzlar O, Kocyigit SE, Aydin AE, Yavuz I, Isik AT. Validation of population-based cutoffs for low muscle mass and strength in a population of Turkish elderly adults. Aging Clin Exp Res. 2020 Sep;32(9):1749-1755. doi: 10.1007/s40520-019-01448-4. Epub 2020 Jan 2. PMID 31898170